CLINICAL TRIAL: NCT03250884
Title: Evaluation of the Performance of a Rapid Pregnancy Diagnostic Test.
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC16_3038
Record Dates: First submitted 2017-08-11; First posted 2017-08-16 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2017-08

CONDITIONS: Pregnancy Related; Diagnostic; Emergencies; Pelvic Pain; Metrorrhagia
MeSH Terms: conditions — Disease; Emergencies; Pelvic Pain; Metrorrhagia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to evaluate the effectiveness of a rapid pregnancy diagnostic test to improve the medical care of patients in emergency room.

DETAILED DESCRIPTION:
The most current gynecological consultations in emergency unit first lead to a pregnancy diagnostic test. The gold standard used is the diagnostic test based on determination of the β-human chorionic gonadotropin concentration. But this assay need time and expect women to wait for hours. A 5-minutes pregnancy diagnostic test has been developed in France. A 62-patients study showed that results obtained with the rapid test were correlated with results obtained with the test based on determination of the β-human chorionic gonadotropin concentration.

The purpose of this study is to evaluate the efficiency of the 5-minutes pregnancy diagnostic test realized in emergency room, in comparison with the blood determination of the β-human chorionic gonadotropin concentration which is only tested in medical laboratory. A little amount of total blood sample used for gold standard test will be used to assess sensibility, specificity, positive or negative predictive values of the rapid pregnancy diagnostic test.

ELIGIBILITY:
Inclusion Criteria:

* Adult women who are in genital activity
* Women who are in emergency unit to consult for metrorrhagia and/or pelvic pains.
* Lack of intrauterine gestational sac determined using endo-vaginal ultrasound
* Women who need a diagnostic test using the β-human chorionic gonadotropin blood test.

Exclusion Criteria:

* Previous pregnancy diagnostic assessed using the β-human chorionic gonadotropin blood test.
* Patients included in an ovarian stimulation program for infertility
* Ectopic gestational sac in which there is an embryo with a cardiac activity determined with ultrasound.
* Patient objecting to participate in the study
* Minor
* Persons subject to major legal protection (safeguarding justice, guardianship, trusteeship), persons deprived of liberty.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnancy test
Study Population: Adult women who come in emergency unit to consult for metrorrhagia and/or pelvic pains and who need a diagnostic test using the β-human chorionic gonadotropin blood test.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-08-30 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Number of diagnostic of pregnancy with the rapid pregnancy diagnostic test in comparison with the number of diagnostic of pregnancy with the blood determination of the β-human chorionic gonadotropin concentration. | 6 months
  Number of diagnostic of pregnancy with the rapid pregnancy diagnostic test in comparison with the number of diagnostic of pregnancy with the blood determination of the β-human chorionic gonadotropin concentration.

SECONDARY OUTCOMES:
Waiting time in emergency unit for patients | 6 months
  Waiting time in emergency unit for patients
Amount of blood tests avoided with the rapid pregnancy diagnostic test | 6 months
  Amount of blood tests avoided with the rapid pregnancy diagnostic test

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Lavoué, Pr, Principal Investigator — Rennes University Hospital
Locations (1):
- Rennes university hospital, Rennes, France